CLINICAL TRIAL: NCT02553018
Title: A National, Randomized, Open-label Study Comparing Compliance and Evolution of Functional Capacity of Patients With Rheumatoid Arthritis Treated With Methotrexate Administered by Auto-injector Versus Administration by Conventional Subcutaneous Injection.
Brief Title: Comparison of Compliance and Evolution of Functional Capacity of Patients With Rheumatoid Arthritis Treated by Methotrexate Either by Auto-injector or by Conventional Sub-cutaneous Syringe
Acronym: Self-i
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MD-112014
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auto-injector of methotrexate (Experimental): The Auto-injector is a disposable, fixed, single dose, auto-injector to be used for Methotrexate (25mg/ml) therapy.
  Dosage form: solution for injection Dosage: 0.3ml contains 7.5mg of Methotrexate, 0.4ml contains the 10.0mg of Methotrexate, 0.6ml contains 15.0 mg of Methotrexate, 0.8ml contains 20.0 mg of Methotrexate, 1.0ml contains 25.0 mg of Methotrexate.
  Frequency: one injection per week Duration: until the end of the study
  Interventions: Drug: Methotrexate
- Pre-filled syringe of methotrexate (Active Comparator): Pre-filled syringes contains a volume of 1 ml with attached injection needle. Dosage form: solution for injection. Dosage: 0.15 ml contains 7.5 mg of methotrexate, 20 ml contains 10 mg of methotrexate, 0.30 ml contains 15 mg of methotrexate, 0.40 ml contains 20 mg of methotrexate, 0.50 ml contains 25 mg of methotrexate disodium.
  Frequency: one injection per week Duration: until the end of the study
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate
  Other Names: Auto-injector of methotrexate; METOJECT

SUMMARY:
The primary objective of the study is to compare, in patients treated with methotrexate injection for rheumatoid arthritis, the compliance and the health assessment questionnaire evolution for the administration by auto-injector versus administration by conventional subcutaneous injection, after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years or over) of either sex.
* With established rheumatoid arthritis diagnosis
* Treated for rheumatoid arthritis by methotrexate (oral or by injection) since at least 3 months regardless of the prior or combined disease modifying treatment, except biotherapies and justifying injection of methotrexate. For the patient treated by oral methotrexate, the switch decided by the rheumatologist is made for either safety, compliance or efficacy issues.
* Agreeing to participate in the study and having dated and signed the informed consent form.

Exclusion Criteria:

* Patients fulfilling one or more of the following exclusion criteria will not be included in the study:

  * Inability of patient to use an auto-injector.
  * Treated with biotherapies.
  * Pregnant or breast-feeding patients
  * Male and female patients with reproductive potential who are not willing to use effective method of contraception (oral contraceptives, intrauterine device, condoms) during study and at least 1 month after the end of the study.
  * Patients with :
* hypersensitivity to methotrexate or to any of the excipients,
* severe hepatic impairment,
* alcohol abuse,
* severe renal impairment,
* pre-existing blood dyscrasias, such as bone marrow hypoplasia, leukopenia, thrombocytopenia or significant anaemia,
* Immunodeficiency,
* serious, acute or chronic infections such as tuberculosis and HIV,
* stomatitis, ulcers of the oral cavity and known active gastrointestinal ulcer disease,
* concurrent vaccination with live vaccines.

  * Association with probenecid, trimethoprim, phenylbutazone.
  * Any other known medical or surgical history, disorder or disease judged by the investigator to be incompatible with the study (such as acute or chronic severe organic disease: hepatic, endocrine, neoplasia, haematological, infectious diseases, severe psychiatric illness, relevant cardiovascular abnormalities, etc…),
  * Inability of patient to understand the study procedures and thus inability to give informed consent.
  * Participation in another clinical study, at the same time as the present study, or during the month following the end of the previous study
  * Ward of court.
  * Patient not covered by the Social Security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Co-primary criteria: observance and health assessment questionnaire | 6 months
  the health assessment questionnaire is completed by the patient at inclusion visit and at the 6 months visit. Compliance with methotrexate treatment will be assessed by the investigator at each visit

SECONDARY OUTCOMES:
quality of life | 6 months
  Patient's quality of life will be assessed using a validated questionnaire. completed by the patient at inclusion and 6 months visits. Change from baseline in questionnaire score will be described.
acceptability | up to 1 year
  The product acceptability will be evaluated by the patient using a specific questionnaire based on several questions related to the patient' opinion, satisfaction and willingness to adopt the product.
preference | 6 months
  Preference will be assessed only for patients receiving auto-injector and pre-filled syringe of methotrexate
Economic | 6 months
  Information on the consumed resources for methotrexate administration will be assessed at 6 months. This information will be further incorporated in a budget impact for the French Sickness Fund

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - SARAUX, Brest
  - HUDRY, Paris

REFERENCES:
- [Derived] Saraux A, Hudry C, Zinovieva E, Herman-Demars H; Self-I Investigators group. Use of Auto-Injector for Methotrexate Subcutaneous Self-Injections: High Satisfaction Level and Good Compliance in SELF-I Study, a Randomized, Open-Label, Parallel Group Study. Rheumatol Ther. 2019 Mar;6(1):47-60. doi: 10.1007/s40744-018-0134-2. Epub 2018 Dec 13. PMID 30547379